CLINICAL TRIAL: NCT04908241
Title: Telerehabilitation With Aims to Improve Lower Extremity Recovery Post-Stroke (TRAIL-RCT): A Randomized Controlled Trial
Brief Title: Telerehabilitation With Aims to Improve Lower Extremity Recovery Post-Stroke (TRAIL-RCT)
Acronym: TRAIL-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Brodie Sakakibara, Assistant Professor, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAIL-RCT
Record Dates: First submitted 2021-05-20; First posted 2021-06-01 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Stroke; Stroke, Ischemic; Stroke Hemorrhagic; Cerebral Injury; Cerebral Infarction; Brain Diseases; Central Nervous System Diseases; Cerebral Vascular Accident; Cerebral Vascular Disorder; Brain Ischemia; Brain Infarction; Cardiovascular Diseases; Infarction
Keywords: Telerehabilitation; Lower Extremity; Self-Management; Education; Secondary Prevention; Stroke; Exercise
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Brain Injuries; Cerebral Infarction; Brain Diseases; Central Nervous System Diseases; Cerebrovascular Disorders; Brain Ischemia; Brain Infarction; Cardiovascular Diseases; Infarction; Motor Activity | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: Following baseline assessment, participants will be randomized into the TRAIL or EDUCATION arm. Following randomization, participants will remain in their allocated group until the completion of the study. A central research coordinator that is not involved in recruitment, assessments or study intervention, will be responsible for randomization of study participants, and will advise the participant and site coordinator of the group allocation. There will be four timepoints where outcome assessments will be conducted, which include baseline (T0), 1-month (T1), 3-months (T2), and 6-months (T3) follow-up.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors will be blinded to participants' group allocation, whereby they will not be involved with delivering the TRAIL or EDUCATION programs. Participants are informed of their group assignment, however they will not know if they are in the experimental or control program, and instructed to withhold it from the assessors to ensure proper blinding and minimize internal bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TRAIL (Experimental): TRAIL is a 4-week progressive exercise and self-management intervention for lower extremity recovery delivered by a trained registered physical therapist, in a 2:1 participant-to-therapist ratio. Each participant grouping will receive two telerehabilitation sessions (60-90 minutes) each week for 4 weeks (total 8-12 hours).
  Interventions: Other: TRAIL
- EDUCATION (Active Comparator): The EDUCATION control arm is a 4-week education program focusing on stroke knowledge and risk factors. It will be delivered by health professionals who have experience working with individuals with stroke, knowledge of chronic disease self-management (e.g. physical or occupational therapists, nurses, kinesiologists), and who have completed study-specific training on the EDUCATION program
  Participants will receive video conferencing sessions with the same schedule and 2:1 participant-to-coach ratio as TRAIL. Each participant grouping will receive two educational telerehabilitation sessions (60-90 minutes) each week for 4 weeks (total 8-12 hours).
  Interventions: Other: EDUCATION

INTERVENTIONS:
Other: TRAIL — Each week has a specific focus for lower extremity rehabilitation:
  Week 1) Building a base: 8 exercises, 10-15 repetitions x 2-3 sets
  Week 2) Increasing repetitions: 8 exercises, 15-20 repetitions x 3 sets
  Week 3) Building exercise tolerance:10 exercises, 15-20 repetitions x 3 sets
  Week 4) Maximizing repetitions: 10 exercises, 30 seconds as many reps as possible x 2 sets
  At the end of the second exercise session each week, the therapist and participants work collaboratively to develop an independent exercise action plan to be completed before the first session of the next week. The self-managed plans includes exercises selected from TRAIL, agreed upon by the participant and therapist, that are safe to perform without therapist oversight. The aims of the exercise action plan are to: i) Add exercise volume without using program resources (e.g., therapist time); and ii) Build capacity for self-management for long-term health and well-being after TRAIL has ended.
  Arms: TRAIL
Other: EDUCATION — EDUCATION has a specific focus on:
  Week 1) What is stroke (e.g., gaining an understanding of the function of the brain, types of stroke and how stroke affects physical function) and introduction to self-management;
  Week 2) What is self-management;
  Week 3) Self-management for post-stroke complications (e.g., activities of daily living);
  Week 4) Self-management for secondary prevention (e.g., blood pressure, diet, medication, stress management).
  Education therapists will be provided with lesson plans and manuals to be circulated with the participants, and will facilitate the educational session through interactive Powerpoint presentations. In addition, participants will be asked to complete 30-60 minutes of educational homework, which will be discussed at the commencement of the following session.
  Arms: EDUCATION

SUMMARY:
The purpose of this study is to compare the effectiveness of a 4-week lower extremity telerehabilitation protocol with aims to improve lower extremity function to a 4-week attention-controlled education program on lower extremity clinical outcomes, quality of life, and healthcare resources utilization among community dwelling adults with stroke across Canada.

DETAILED DESCRIPTION:
With an aging population, and survival rates now at 83% in Canada, the number of stroke survivors is expected to reach 720,000 by 2038. While 90% of individuals with stroke return to independent community living, 80% report residual motor impairment, such as loss or limitation in motor control, or mobility limitation. These limitations have profound effects on the ability to perform everyday activities and are associated with substantial economic strain on the healthcare system. Thus, a primary focus of stroke rehabilitation is on the recovery of motor function, walking and balance, using exercise via physical therapy.

The rapid growth in Internet use and personal mobile devices has opened an array of possibilities for stroke survivors to remotely access specialized rehabilitation from their homes and communities (i.e., telerehabilitation). Telerehabilitation interventions have been used effectively for check-in sessions, education, and counselling after stroke, but knowledge of the effectiveness of using telerehabilitation for the delivery of exercise interventions for lower extremity recovery is limited.

The investigators developed the TeleRehabilitation with Aims to Improve Lower Extremity Recovery Post-Stroke (TRAIL) to address the unmet needs for lower extremity rehabilitation after stroke, and the need for accessible rehabilitation in the face of the COVID-19 pandemic. TRAIL is an exercise program designed to promote lower extremity recovery using technology with real-time therapist instruction and guidance. The investigators recently conducted a proof-of-concept, single-group feasibility study of TRAIL (TRAIL-PROOF). From TRAIL-PROOF, there were have no reports of serious adverse events and 100% retention of participants. Preliminary analysis of 32 individuals completed also suggest improvements in the clinical outcomes, including increased lower extremity strength, functional balance, and balance self-efficacy. Thus, from TRAIL-PROOF, it is evident that the TRAIL protocol has potential to improve lower extremity function among community-dwelling adults with stroke experiencing lower extremity impairment. The investigators now propose a full-scaled randomized controlled trial to further study the TRAIL program (TRAIL-RCT).

The objectives for TRAIL-RCT are as follows:

1. The primary objective is to compare functional mobility (Timed Up and Go, primary clinical outcome) after 4 weeks of TRAIL to a 4-week attention-controlled education program (EDUCATION) in individuals ≤12 months post-stroke;
2. The secondary objective is to compare the 4-week TRAIL and EDUCATION programs on secondary outcomes of:

   1. Lower extremity strength (30-Second Sit-to Stand test);
   2. Functional balance (Tandem Stand and Functional Reach);
   3. Motor impairment (Virtual Fugl-Meyer Assessment);
   4. Balance self-efficacy (Activities-specific Balance Confidence Scale);
3. The tertiary objective is to compare the 4-week TRAIL and EDUCATION programs on health economic outcomes:

   1. Health-related quality of life (Stroke Impact Scale, EuroQol-5D-5 Level); and
   2. Health resources and costs (Health Resource Utilization Questionnaire)
4. The quaternary objective is to evaluate the feasibility of a subsequent larger multisite implementation stepped wedge randomized trial of TRAIL using pre-specified criteria related to process, resources, management, and scientific indicators.

It is hypothesized that:

The primary hypothesis is that the 4-week TRAIL program will lead to greater improvement in functional mobility, as measured by the Timed Up and Go, compared to the 4-week EDUCATION program in individuals ≤12 months post-stroke (Objective 1, primary clinical outcome).

The investigators also anticipate that greater improvements will be observed in the secondary clinical outcomes, in the areas of lower extremity muscle strength, motor impairment, functional balance, and balance self-efficacy, following TRAIL compared to EDUCATION (Objective 2).

The tertiary hypothesis is that the TRAIL intervention will demonstrate superior health economic outcomes compared to the EDUCATION group (Objective 3).

The quaternary hypothesis is that the protocol will demonstrate sufficient feasibility (e.g., rates of recruitment/retention, treatment fidelity and adherence, safety, treatment effects) to support a subsequent larger multi-site implementation stepped wedge randomized controlled trial (Objective 4).

ELIGIBILITY:
Inclusion Criteria:

* ≥19 years of age, ≤12 months post-stroke with lower extremity hemiparesis
* Able to walk ≥10 meters with or without a gait aid and without physical assistance of another person
* Can tolerate 50 minutes of activity (including rest breaks)
* Has cognitive-communicative ability to participate, per clinical judgement
* Able to provide consent
* Has a caregiver, friend, or family member available to provide physical support during the assessment sessions

Exclusion Criteria:

* Currently participating in formal in- or out-patient stroke rehabilitation focusing on lower extremity training
* Living in long-term care
* Severe vision or hearing loss
* Significant musculoskeletal or other neurological conditions
* Not medically stable
* Comorbidities (e.g. limb amputation), pain or other symptoms that significantly impact lower extremity function
* Planned surgery that would preclude or affect participation in the protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Timed Up and Go (TUG) at 4 weeks | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Performance walking test to assess functional mobility

SECONDARY OUTCOMES:
Stroke Impact Scale (SIS) | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Stroke specific, self-reported health status measure. There are 8 domains assessed in this version and each item is rated using a 5-point Likert scale. The participant rates his/her difficulty completing the task from 1 to 5, where lower scores mean greater difficulty to complete the item.
Activities-Specific Balance (ABC) Scale | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Self-reported questionnaire measuring self-efficacy in performing activities without losing balance. The ABC Scale consists of 16 questions that require the participant to rate their confidence in performing the activity from 0% to 100%, where higher percentages indicate greater self-efficacy
Functional Reach | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Performance measure to assess balance through maximal forward reach (in cm) from a fixed base
Modified Virtual Fugl-Meyer Assessment | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Performance measure to assess lower extremity impairment
30 second Sit to Stand | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Performance measure used to assess lower extremity strength
Health Resource Utilization Questionnaire | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Health care utilization calculated by assessing health professional visits, admissions to hospital, laboratory tests/ investigations, and use of medications
Health-related quality of life (EuroQol-5D-5 Level) | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  A generic preference-based utility instrument composed of 5 domains of health (mobility, self-care, usual activities, pain, anxiety/depression), each with 5 levels (1=no problems, 5=major problems), which is often used to calculate cost-utility
Tandem Stand | Baseline, Post-Intervention (immediately following 4 weeks of intervention), 3-months, 6-months
  Performance measure to assess balance through holding a tandem stance position (up to 10 seconds; alternate positions: semi-tandem or feet together

OTHER OUTCOMES:
Feasibility Indicator: Recruitment Rate | Study Completion (Post-Intervention, immediately following study completion)
  Number of participants recruited
Feasibility Indicator: Retention Rate | Study Completion (Post-Intervention, immediately following study completion)
  Number of participants with post-intervention data
Feasibility Indicator: Perceived Benefit of Telerehabilitation | Post-Intervention (immediately following 4 weeks of intervention)
  Satisfaction survey administered at the end of post-intervention visit
Feasibility Indicator: Treatment Fidelity | Post-Intervention (immediately following 4 weeks of intervention)
  Percentage of telerehabilitation sessions attended, exercise completed during telerehabilitation sessions, and self-management sessions completed
Feasibility Indicator: Blinding of Outcome Assessors | Study Completion (Post-Intervention, immediately following study completion)
  Percentage of outcome assessors remaining blinded to group allocation throughout duration of study
Feasibility Indicator: Appropriateness of Randomization Process | Study Completion (Post-Intervention, immediately following study completion)
  Number of participants per group and baseline differences in outcomes between groups
  Baseline differences between groups
Feasibility Indicator: Number of Participants Excluded based on Eligibility Criteria | Study Completion (Post-Intervention, immediately following study completion)
  Number of individuals excluded from potential participant list (referrals from inpatient stroke rehabilitation and community outreach)
Feasibility Indicator: Participant and Assessor Burden | Study Completion (Post-Intervention, immediately following study completion)
  Duration (measured in minutes) to complete the assessments.
Feasibility Indicator: Participant Burden | Study Completion (Post-Intervention, immediately following study completion)
  Percentages of participants with pre- and post-assessments
Feasibility Indicator: Ease of Using Equipment | Study Completion (Post-Intervention, immediately following study completion)
  Downtime due to technical issues of tablet and video-conferencing platform (measured in minutes)
Feasibility Indicator: Safety | Study Completion (Post-Intervention, immediately following study completion)
  Number of adverse events from the program sessions or assessments
Feasibility Indicator: Processing Time | Study Completion (Post-Intervention, immediately following study completion)
  Time from initial contact to enrolment
GENESIS-PRAXY Questionnaire | Baseline Assessment
  Questionnaire used to assess gender-related measures encompassing gender roles, relations and identity. A composite score is calculated to determine whether an individual has primarily masculine, neutral or feminine gender characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Brodie Sakakibara, PhD, Principal Investigator — University of British Columbia; Ada Tang, PhD, Principal Investigator — McMaster University
Locations (5):
- Canada (5):
  - University of British Columbia, Vancouver, British Columbia
  - Dalhousie University, Nova Scotia, Halifax
  - Riverview Health Centre, Winnipeg, Manitoba
  - Parkwood Institute, London, Ontario
  - University Health Network, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
The anonymized data collected during the study, the trial protocol, statistical analysis plan, and informed consent form will be shared with qualified researchers engaging in independent scientific research, upon request to the research team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After the study end.
Access Criteria: Please contact the research team.

REFERENCES:
- [Derived] Sakakibara BM, Wiley E, Barclay R, Bayley M, Davis JC, Eng JJ, Harris A, Inness EL, MacKay-Lyons M, Monaghan J, Pollock C, Pooyania S, Schneeberg A, Teasell R, Yao J, Tang A. TeleRehabilitation with Aims to Improve Lower extremity recovery in community-dwelling individuals who have had a stroke: protocol for a multisite, parallel group, assessor-blinded, randomised attention-controlled trial. BMJ Open. 2023 Jul 19;13(7):e076723. doi: 10.1136/bmjopen-2023-076723. PMID 37474180